CLINICAL TRIAL: NCT02888587
Title: The Innervation of Human Gut Sensory Epithelial Cells
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00075870
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Organoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — To obtain endoscopic and colonoscopic biopsies to harvest and culture intestinal crypts from human tissue to produce organoids. These organoids will be used to study the biology of innervated sensory epithelial cells.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: no gastrointestinal symptoms
- Symptomatic group: Patients with Visceral hypersensitivity

SUMMARY:
The study has two objectives:

1. To obtain endoscopic and colonoscopic biopsies to harvest and culture intestinal crypts from human tissue to produce organoids. These organoids will be used to study the biology of innervated sensory epithelial cells.
2. to collect subject data relating to clinical management and demographic characteristics of patients undergoing upper endoscopy or colonoscopy to learn the mechanisms behind visceral hypersensitivity, and neurodegenerative diseases that may arise in the gut.

DETAILED DESCRIPTION:
Throughout the gastrointestinal tract there are specialized sensory epithelial cells that recognize stimuli from nutrients and bacteria. These cells have been traditionally known for their endocrine function. However, it was recently discovered using mouse models that these cells receive synaptic inputs from enteric and peripheral neurons, such as those with cell bodies in dorsal root ganglia or the vagal nodose.

This finding opened a few possibilities, including the following: 1) sensory function of the gastrointestinal tract is modulated by neural activity; 2) gut bacteria influences brain function through a direct neural circuit; and 3) viruses that preferentially infect neurons access the central nervous system through this neural circuit [1,2]. To translate findings in animal models to humans, the investigator must test the hypotheses in which the physiology of gut sensory epithelial cells resembles that of humans.

Visceral hypersensitivity is a core symptom for several gastrointestinal and brain behavior disorders, including irritable bowel syndrome, autism and anorexia. Unfortunately, the basic mechanisms of sensory processing in the wall of the gut are non-existent. This lack of knowledge precludes the development of therapeutic strategies to treat disorders linked to visceral hypersensitivity. The investigator's efforts to translate animal research into human models will be a foundation to develop target therapies for visceral hypersensitivity.

Today, it is possible to derive organoids from intestinal crypts harvested from human intestinal or colonic tissue. The organoids have all epithelial cell types, including gut sensory cells. Here, the investigator's goal is to use de-identified human tissues to culture intestinal organoids in the laboratory, and use it as a platform to study the biology of innervated sensory epithelial cells. This work is significant because it will open the possibility to learn the mechanisms behind visceral sensation and neurodegenerative diseases that may arise in the gut.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing either endoscopy OR colonoscopy OR both procedures will be eligible for inclusion in this study.
* adult males and females 18 years of age or older who have been seen by the GI clinic or who have been scheduled for direct-to-procedure appointment in the GI clinic.

Exclusion Criteria:

* Subjects who are not competent to give consent
* Males and females under 18 years of age
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be identified as they are seen by the GI group during scheduled appointments, laboratory tests or endoscopic or operative procedures. All patients undergoing either endoscopy OR colonoscopy OR both procedures will be eligible for inclusion in this study
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Expression of sensory receptors in enteroendocrine cells | 4 years
  Organoids are expected to contain enteroendocrine cells. We will use electrophysiology to measure the electrical excitability of these cells. In enteroendocrine cells from patients with a visceral hypersensitivity diagnosis is expected that cells will fire action potentials at a significantly lower threshold. These results will be correlated with RNA sequencing analysis to study the expression of sensory receptors in enteroendocrine cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data stays at Duke Medical Center.